CLINICAL TRIAL: NCT00676767
Title: Resistant Starch Type 4 on the Glycemic Response in Older Adults
Brief Title: Resistant Starch on Glycemic Response in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: MGP Ingredients, Inc. (Industry)
Responsible Party: Mark D. Haub, Ph.D., Associate Professor, Kansas State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: KSU-HML-RSt1
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Hyperglycemia
Keywords: Aging; Diabetes; Diet; Fiber
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Dietary Supplement: Resistant Starch Type 4
- 2 (Active Comparator)
  Interventions: Dietary Supplement: Dextrose
- 3 (Placebo Comparator)
  Interventions: Dietary Supplement: Puffed wheat

INTERVENTIONS:
Dietary Supplement: Resistant Starch Type 4
  Arms: 1
Dietary Supplement: Dextrose
  Arms: 2
Dietary Supplement: Puffed wheat
  Arms: 3

SUMMARY:
The purpose of this study was to determine how blood glucose changes after eating energy bars containing resistant starch type 4 compared with bars made with puffed wheat in healthy older adults.

DETAILED DESCRIPTION:
To measure the blood glucose response, we collected blood samples before eating and 15, 30, 45, 60, 90 and 120 minutes after eating each bar. The incremental area under the curve was used to calculate glycemic index.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy (not diagnosed with disease)
* Over 60 years of age

Exclusion Criteria:

* Diagnosed with diabetes or other metabolic disorder
* Allergies to wheat
* Non-smokers

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Glycemic Response | 2-hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Haub, Ph.D, Principal Investigator — Kansas State University
Locations (1):
- Human Metabolism Laboratory, Manhattan, Kansas, United States